CLINICAL TRIAL: NCT04431596
Title: Computational Initiative for Performance Monitoring: Military Alerting System for Monitoring Body Temperature During Active Cooling
Brief Title: Military Alerting System for Monitoring Body Temperature During Active Cooling
Acronym: MAMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Biotechnology High Performance Computing Software Applications Institute (Unknown)
Responsible Party: Principal Investigator, Douglas J Casa, Professor, University of Connecticut
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H20-0010
Record Dates: First submitted 2020-05-27; First posted 2020-06-16 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Intervention Model Description: Participants receive three cooling treatments on separate study visits: 1) passive cooling 2) mist-fan cooling and 3) forearm immersion cooling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooling (Active Comparator): Participants will be actively cooled during rest breaks.
  Interventions: Device: Forearm cooling; Other: Mist-fan cooling
- No Cooling (No Intervention): Participants will participant in "passive cooling" where they sit in a chair during rest.

INTERVENTIONS:
Device: Forearm cooling — forearm immersion will be performed for active cooling assessment.
  Arms: Cooling
Other: Mist-fan cooling — A mist-fan will be placed in front of the participant for active cooling.
  Arms: Cooling

SUMMARY:
BHSAI is developing a computational system that provides early alerts of a rise in core body temperature to help reduce the risk of heat injury in the field and during training. The goal of the body temperature alerting system is to use it during rest, exercise in the heat and during body cooling. Using this system during cooling will allow healthcare professionals and military personnel monitor core temperature to ensure cooling is effective (and prevent hypothermia). Therefore, the primary purpose of this investigation is to validate a body temperature alerting system using physiological responses that occur during rest, exercise in the heat and during body cooling. Multiple cooling modalities will be validated. The effectiveness of each cooling modality (passive cooling, mist-fan cooling, hand/forearm immersion) on physiological variables after exercise in the heat will be assessed. Lastly, subject characteristics (demographic and anthropometric characteristics) will be examined to examine their effect on physiological variables during exercise in the heat and during body cooling with each cooling modality.

DETAILED DESCRIPTION:
The study will be completed in the following timeline:

Visit 1: Baseline and VO2max Testing Visit 2-4: Trial 1, 2 and 3

Visit specific information is described below, however, specific data collection protocols for dependent variables and procedures are included below the description of the study design.

Visit 1: Baseline and VO2max Testing

Participants who are approved to participate will be scheduled for a baseline and VO2max testing day. Upon arrival to the lab, subjects will provide a urine sample in a clean urine cup. Urine specific gravity and urine color will be assessed. Nude body mass will be also be recorded. Privacy will be afforded for each participant while obtaining body mass measures by taking measurements with the participant alone in a private room behind a solid, closed door, and the research reading the scale outside of the room. Participants will only be permitted to continue to the VO2max test if the euhydrated criteria of a urine specific gravity (USG) <1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the subject will be asked to drink 500 mL of water to ensure proper hydration status. Height will be measured with a tape measure on Visit 1. Percent body fat will be calculated using a 7-site evaluation of skin fold thickness using skin fold calipers. A researcher will use appropriate grasping technique to measure skin fold thickness on the chest, iliac, tricep, calf, shoulder, abdomen, and thigh. This will take less than 5 minutes to complete. This information will be used to describe the subject demographics. Participants will also be asked to complete a maximal oxygen uptake (VO2max) test on a treadmill in a thermoneutral environment. This test will provide aerobic fitness levels of the participants. This visit will take approximately 1-2 hours.

Visit 2-3: Trials 1, 2, 3

Participant numbers will be randomly assigned, and trials will be ordered with a random number generator and assigned to a participant number. These orders will be counterbalanced between participants to ensure that there is not an order effect, and each participant will complete three trials as part of the study. Participants will be allowed to make-up trial visits if they are sick, suffer an injury or do not meet hydration requirements. Participants will be asked if they have a current illness or taking medications to determine whether they can complete the exercise trial. The participant's visit will be rescheduled if they have a fever, current illness or taking medications that influence body temperature.

Participants will complete three trials on three separate days in a randomized counter balanced order:

Trial Cooling Intervention

1. Passive Cooling
2. Mist-fan Cooling
3. Forearm Immersion

The exercise protocol and recovery portions of this study will be conducted in a climatic chamber with ambient temperature approximately 30-40C and relative humidity at approximately 30-70%. Participants will drink ad libitum throughout the exercise trial.

Upon arrival to the lab, participants will be asked to indicate if they have consumed alcohol or caffeine in the last 24 hours and 12 hours, respectively. They will not be asked to specify exactly what they have consumed, but if they provide a positive indication, their trial will be rescheduled for another day. Participants will provide a small urine sample in a clean urine cup, and a nude body mass will be measured. Upon arrival to the lab, hydration status will be assessed by urine specific gravity, nude body mass and urine color. Participants will only be permitted to continue to the exercise trial if the euhydrated criteria of a urine specific gravity (USG) <1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the subject will be asked to drink 500 mL of water to ensure proper hydration status. Participants will be given instructions at the prior visit about how to obtain desired hydration status for the upcoming trial. Participants will insert a rectal probe and wear a heart rate monitor strap. Additionally, participants will wear 7-site skin temperature sensors. Researchers will apply the skin temperature sensors with medical tape to the participants' chest, upper arm, thigh, neck, abdomen, thigh, back, and calf. The participants will also be asked to complete a subjective sleep questionnaire upon arriving to the lab. Participants will wear a battle dress uniform (BDU) during all exercise and rest blocks. Three BDU sizes for the blouse and pants (small, medium, large) will be available for the participants. A belt will be used to ensure the BDU fits appropriately. Participants will not be able to keep the BDU- BDUs will be washed (according to manufacturer's instructions) and re-used for participants. BDU manufacturer's instructions is identical to standard washing cycle (detergent and washing machine dry). Participants will wear the wrist-based devices (provided by BHSAI) on their non-dominant arm throughout the testing. The wrist device must be placed approximately 1-inch proximal to the wrist and be fitted snuggly for accurate heart-rate measurements. The wrist device is used to estimate heart rate using infrared technology. The wrist device estimates of heart rate will be compared to the polar heart rate monitor (gold standard). The body alerting system uses heart rate from the wrist device and the environmental conditions to estimate body temperature. The sponsor of the study will use rectal temperature and the 7-site skin temperature sensors to alter the algorithm (not in real time- from the collected data) to better estimate body temperature. The future goal is to have the body alerting system imbedded in the watch.

Participants will enter the environmental chamber and sit for 30 minutes to become equilibrated. The environmental chamber will be set to 36C ambient temperature, 30% relative humidity After baseline measures of heart rate, rectal temperature, participants will complete the perceptual indices. Participants will also complete an environmental symptoms questionnaire (ESQ).

The trial will consist of three, 50-minute intervals of walking and running at approximately 30-50% of VO2max and 60-80% of VO2max, respectively. Each 50-minute exercise block with be followed by a 30-minute break where cooling will occur. Participants will be allowed to drink ad libitum throughout the exercise trial. The participant will be cooled for approximately 30 minutes with their assigned cooling modality. Rectal temperature, skin temperature, heart rate, perceptual measures, and mood will be collected at various time points before, during, and after exercise and cooling.

Passive Cooling: Participants will be asked to sit in a chair in the climate chamber for passive cooling.

Mist-fan cooling: A mist-fan will be placed in front of the participant during mist-fan cooling. Participants will be asked to roll up their BDU sleeves to increase skin surface area. The temperature of the mist and wind speed of the fan will be recorded.

Forearm immersion: The participant will place their forearm in approximately 20C water during forearm immersion.

Data collection will be divided into two separate phases. A pilot study will be first conducted in which the first two participants will complete all study laboratory visits. Data from those trials will be shared with the sponsor for review before continuation of data collection.

Participants will undergo the same procedures for the pilot testing as regular testing. Pilot testing data will be included in the dataset. Following approval from the sponsor, data collection will resume. Each trial will be approximately 4-5 hours.

All devices will be properly cleaned according to manufacturer's instruction prior to use by other participants.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender man between the ages of 18-35 years
* been cleared by the medical monitor for this study
* VO2max > 45ml/kg/min

Exclusion Criteria:

* Have a current musculoskeletal injury that would limit their physical activity or preclude the participant from walking, jogging, running, sprinting, or cutting.
* Chronic health problems that affect your ability to thermoregulate (disorders affecting the liver, kidneys or the ability to sweat normally)
* Fever or current illness at the time of testing
* History of cardiovascular, metabolic, or respiratory disease
* Current musculoskeletal injury that limits their physical activity
* Currently taking a medication that is known to influence body temperature (amphetamines, antihypertensives, anticholinergics, acetaminophen, diuretics, NSAIDs, aspirin)
* Identify as cisgender woman, transgender man or transgender woman
* Have a history of heat related illness

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Change in Rectal Temperature | Measured continuously for 50 min exercise block 1, 30 min cooling period block 1, 50 min exercise block 2, 30 min cooling period block 2, 50 min exercise block 3, 30 min cooling period block 3 (total 240 minutes)
  Rectal thermometer will be self-inserted by participant to assess core temperature
Change in Mean Skin Temperature | Measured continuously for 50 min exercise block 1, 30 min cooling period block 1, 50 min exercise block 2, 30 min cooling period block 2, 50 min exercise block 3, 30 min cooling period block 3 (total 240 minutes)
  7 skin temperature sensors will be placed on the subject (neck, chest, shoulder,back, abdomen, thigh, calf)
Change in Heart Rate | Measured continuously for 50 min exercise block 1, 30 min cooling period block 1, 50 min exercise block 2, 30 min cooling period block 2, 50 min exercise block 3, 30 min cooling period block 3 (total 240 minutes)
  A heart rate monitor will be worn by participant throughout exercise/cooling protocol
Change in Rating of Perceived Exertion (RPE) | Measured every 10 minutes during 50 min exercise block 1, 30 min cooling period block 1, 50 min exercise block 2, 30 min cooling period block 2, 50 min exercise block 3, 30 min cooling period block 3 (total 240 minutes)
  6-20 scale that indicates how hard the participant feels they are working. 6 represents rest and 20 represents maximal exertion. A high score indicates more perceived exertion.
Change in Thermal Sensation (TS) | Measured every 10 minutes during 50 min exercise block 1, 30 min cooling period block 1, 50 min exercise block 2, 30 min cooling period block 2, 50 min exercise block 3, 30 min cooling period block 3 (total 240 minutes)
  0-8 Scale (cold to hot) that indicated how cold or hot the participate feels. 0 = extremely cold, 8 = extremely hot.
Change in Perception of Fatigue | Measured every 10 minutes during 50 min exercise block 1, 30 min cooling period block 1, 50 min exercise block 2, 30 min cooling period block 2, 50 min exercise block 3, 30 min cooling period block 3 (total 240 minutes)
  0-10 (no fatigue to extreme fatigue) Scale that indicates how fatigued the participate feels. High score indicates more fatigue (negative outcome).
Change in Perception of Thirst | Measured every 10 minutes during 50 min exercise block 1, 30 min cooling period block 1, 50 min exercise block 2, 30 min cooling period block 2, 50 min exercise block 3, 30 min cooling period block 3 (total 240 minutes)
  0-9 (no thirst to extreme thirst) Scale that indicates how thirsty the subject feels. A higher score is considered a negative outcome.
Environmental Symptoms | Before the start of exercise block 1
  An environmental symptoms questionnaire to indicate they feel (hot, lethargic, irritable)
Environmental Symptoms | After the 30 min cooling period in block 3
  An environmental symptoms questionnaire to indicate they feel (hot, lethargic, irritable)

SECONDARY OUTCOMES:
POMS | Immediately before exercise block 1
  Questionnaire that indicates the current mood of the participant
POMS | Immediately following cooling period in block 1
  Questionnaire that indicates the current mood of the participant
POMS | Immediately following cooling period in block 2
  Questionnaire that indicates the current mood of the participant
POMS | Immediately following cooling period in block 3
  Questionnaire that indicates the current mood of the participant
Heart Rate Variability | Measured continuously for 50 min exercise block 1, 30 min cooling period block 1, 50 min exercise block 2, 30 min cooling period block 2, 50 min exercise block 3, 30 min cooling period block 3 (total 240 minutes), then for 5 minutes 24 hours after
  The device used to collect HR (polar) will be used to collect heart rate variability
Digits Backwards | immediately before exercise block 1
  A cognitive assessment where participants are asked to repeat a series of numbers backwards, the numbers will be read out loud by the researcher.
Digits Backwards | immediately following cooling block 2
  A cognitive assessment where participants are asked to repeat a series of numbers backwards, the numbers will be read out loud by the researcher.
Digits Backwards | immediately following cooling block 3
  A cognitive assessment where participants are asked to repeat a series of numbers backwards, the numbers will be read out loud by the researcher.
Purdue Peg Board test | immediately before exercise block 1
  A hand dexterity assessment that measures how quickly the participant can place a pins into a pegboard (left and right hand)
Purdue Peg Board test | immediately after cooling block 2
  A hand dexterity assessment that measures how quickly the participant can place a pins into a pegboard (left and right hand)
Purdue Peg Board test | immediately after cooling block 3
  A hand dexterity assessment that measures how quickly the participant can place a pins into a pegboard (left and right hand)
Psychomotor Vigilance Test | immediately before exercise block 1
  a reaction time test (on a samsung phone) where participants are asked to press the number numbers as quickly as they can
Psychomotor Vigilance Test | immediately after cooling block 2
  a reaction time test (on a samsung phone) where participants are asked to press the number numbers as quickly as they can
Psychomotor Vigilance Test | immediately after cooling block 3
  a reaction time test (on a samsung phone) where participants are asked to press the number numbers as quickly as they can
Digit Vigilance Test | immediately before exercise block 1
  Participants are given 2 pages of numbers and are asked to cross out all the 6's (or 9's) as quickly and accurately as they can.
Digit Vigilance Test | immediately after cooling block 2
  Participants are given 2 pages of numbers and are asked to cross out all the 6's (or 9's) as quickly and accurately as they can.
Digit Vigilance Test | immediately after cooling block 3
  Participants are given 2 pages of numbers and are asked to cross out all the 6's (or 9's) as quickly and accurately as they can.
Trial Making Test | immediately before exercise block 1
  Participants are asked to connect as series of numbers and letters together (using a pencil)
Trial Making Test | immediately after cooling block 2
  Participants are asked to connect as series of numbers and letters together (using a pencil)
Trial Making Test | immediately after cooling block 3
  Participants are asked to connect as series of numbers and letters together (using a pencil)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Casa, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Gampel Pavilion, Storrs, Connecticut, United States